CLINICAL TRIAL: NCT02841618
Title: The Healthy Cookie Study: Understanding How Healthy Cookies Affect Fat in the Blood,
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Martha Belury, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015H0209
Record Dates: First submitted 2016-07-15; First posted 2016-07-22 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Healthy Adults

STUDY DESIGN:
Intervention Model Description: Two Phases:
  Phase 1: Single arm, grapeseed oil cookie (N=39 adults) Phase 2: Triple masked, grapeseed or safflower oil cookie (N=84 adults)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- High Linoleic Acid Healthy Cookies (Experimental): High Linoleic Acid Healthy Cookies (10g grapeseed oil) 1 per day for 2 weeks Phase 1: N=39 adults single arm Phase 2: N=42 adults
  Interventions: Other: High Linoleic Acid Healthy Cookies
- High Oleic Acid Healthy Cookies (Placebo Comparator): High Oleic Acid Healthy Cookies (10g safflower oil) 1 per day for 2 weeks Matched for Phase 2: N=42 adults
  Interventions: Other: High Oleic Acid Healthy Cookies

INTERVENTIONS:
Other: High Linoleic Acid Healthy Cookies
  Arms: High Linoleic Acid Healthy Cookies
Other: High Oleic Acid Healthy Cookies
  Arms: High Oleic Acid Healthy Cookies

SUMMARY:
The purpose of this study is to understand how consuming healthy cookies every day for two weeks will affect different types of fat in the blood. Specifically, the overall goal of this study is to find out if the healthy cookies can increase a polyunsaturated fat called linoleic acid in plasma, red blood cells and white blood cells.

DETAILED DESCRIPTION:
Overall, linoleic acid has many health benefits including altering body composition and energy metabolism, possibly through its impact on cardiolipin. It is therefore imperative to develop foods products that allow for Americans to easily increase their intake of linoleic acid. It's also important to understand the mechanism in which linoleic acid exerts these positive health effects, particularly in states of muscle mass and quality loss associated with mitochondria dysfunction.

The investigators plan to test the central hypothesis and accomplish the overall objective of this research by pursuing the following three specific aims

Aim 1: To determine the extent to which cookies, made with grapeseed oil , increase linoleic acid in plasma, red blood cells (RBCs), and peripheral blood mononuclear cells (PBMCs) fraction of blood after two weeks consumption

Aim 2: To determine the extent to which cookies, made with grapeseed oil, increase cardiolipin and linoleic acid content of cardiolipin in PBMCs after two weeks of consumption

Aim 3: To determine and compare the acceptability of consuming cookies made with grapeseed oil or high oleic safflower oil every day for two weeks

ELIGIBILITY:
Inclusion Criteria:

* Nonsmokers

Exclusion Criteria:

* Current or previous diagnosis of diabetes, heart (including stroke or heart attack), kidney, liver or circulatory diseases and/or current treatment for cancer.
* Gastrointestinal diseases or disorders (including pancreatic) or gastric bypass surgery
* Food Allergy or Intolerance & Bee allergy
* Any dietary restriction where consumption of these healthy cookies or any ingredient would be contraindicated
* Use of medications where consuming the healthy cookies would be contraindicated
* Use of supplements/oils high in linoleic acid in the past 4 weeks prior to enrolling
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in fasting fatty acid levels | Baseline through Week 02
  Linoleic acid content of fasting blood samples
Changes in cardiolipin | Baseline through Week 02
  Cardiolipin content in fasting blood samples
Acceptability of Cookies | Baseline through Week 02
  9-point sensory evaluation of healthy cookies

SECONDARY OUTCOMES:
Correlation of linoleic acid in the blood with body strength | Baseline through Week 02
  grip strength measurement
Correlation of linoleic acid in the blood with body movement | Baseline through Week 02
  gait speed measurement
Correlation of linoleic acid in blood with body size | Baseline through Week 02
  Body Mass Index measurement
Correlation of linoleic acid in blood with body shape | Baseline through Week 02
  Abdominal thickness measurement
Correlation of linoleic acid in blood with sleep | Baseline through Week 02
  Sleeping questionnaire
Correlation of linoleic acid in blood with physical activity | Baseline through Week 02
  Physical Activity questionnaire
Correlation of fatty acids in blood with diet | Baseline through Week 02
  omega-3 fat intake questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Human Nutrition Laboratory, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No